CLINICAL TRIAL: NCT06174831
Title: Study of a Series of Patients Treated for Retrograde Cricopharyngeal Muscle Dysfunction Syndrome
Acronym: R-CPD-Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8782
Record Dates: First submitted 2023-10-23; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-10

CONDITIONS: Deglutition Disorders
Keywords: Deglutition Disorders; Dysphagia; cricopharyngeus muscle; Circular sphincter; Esophagus; Botulinum toxin
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
R-CPD syndrome (Retrograde Cricopharyngeal Dysfunction syndrome) is an inability to burp.

It is a syndrome whose diagnosis is clinical, and for which there is effective treatment. Recently treated in the United States (first publication in 2019), this syndrome affects many patients in France and is currently unknown.

This study concerns a series of patients treated at the University Hospitals of Strasbourg for a syndrome of retrograde dysfunction of the cricopharyngeus muscle having been treated by injection of botulinum toxin into the cricopharyngeus muscle.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject treated by injection of botulinum toxin into the cricopharyngeal muscle after having had a diagnosis of R-CPD in consultation between January 1, 2022 and December 31, 2022
* Subject not opposing the reuse of their data for the purposes of this research.

Exclusion Criteria:

* Subject having expressed opposition to participating in the study,
* Subject under judicial protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major Subject treated by injection of botulinum toxin into the cricopharyngeal muscle after having had a diagnosis of R-CPD in consultation between January 1, 2022 and December 31, 2022
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01-19 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the characteristics of a series of patients treated for dysphagia syndrome | Through study completion, an average of 2 months
  Retrospective study of medical files of patients treated in HUS between January 1, 2022 and December 31, 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-faciale - CHU de Strasbourg - France, Strasbourg, France